CLINICAL TRIAL: NCT05814731
Title: A Randomized Controlled Study on the Efficacy and Safety of MA-BUCY2 Protocol in the Conditioning of Haploidentical Stem Cell Transplantation in Patients With High-risk Acute Myeloid Leukemia
Brief Title: Study on the Efficacy and Safety of MA-BUCY2 Conditioning in High-risk AML Patients Underwent Haplo-HSCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2022SJ-XK005
Record Dates: First submitted 2023-02-22; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Haploidentical Stem Cell Transplantation; Conditioning
MeSH Terms: interventions — Cytarabine; Busulfan; Cyclophosphamide; Semustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MA-BUCY2 (Experimental): Mitoxantrone liposome 20mg/m2，ivgtt，d-11 ；Ara-C 4g/m2.d ，ivgtt，d-10- -9； BU 0.8 mg/kg q6h，ivgtt，d-8- -6； CTX 1.8 g/m2.d ，ivgtt，d-5- -4； me-CCNU 250 mg/m2，p.o，d-3； ATG 2.5 mg/Kg.d，d-5 -2；
  Interventions: Drug: MA-BUCY2
- BUCY2 (Active Comparator): Ara-C 4g/m2.d ，ivgtt，d-10- -9； BU 0.8 mg/kg q6h，ivgtt，d-8- -6； CTX 1.8 g/m2.d ，ivgtt，d-5- -4； me-CCNU 250 mg/m2，p.o，d-3； ATG 2.5 mg/Kg.d，d-5 -2；
  Interventions: Drug: BUCY2

INTERVENTIONS:
Drug: MA-BUCY2 — Mitoxantrone liposome 20mg/m2，ivgtt，d-11 ；Ara-C 4g/m2.d ，ivgtt，d-10- -9； BU 0.8 mg/kg q6h，ivgtt，d-8- -6； CTX 1.8 g/m2.d ，ivgtt，d-5- -4； me-CCNU 250 mg/m2，p.o，d-3； ATG 2.5 mg/Kg.d，d-5 -2
  Other Names: Mitoxantrone liposome; cytarabine; busulfan; cyclophosphamide; semustine; anti-thymocyte immunoglobulin
  Arms: MA-BUCY2
Drug: BUCY2 — Ara-C 4g/m2.d ，ivgtt，d-10- -9； BU 0.8 mg/kg q6h，ivgtt，d-8- -6； CTX 1.8 g/m2.d ，ivgtt，d-5- -4； me-CCNU 250 mg/m2，p.o，d-3； ATG 2.5 mg/Kg.d，d-5 -2
  Other Names: Cytarabine; busulfan; cyclophosphamide; semustine; anti-thymocyte immunoglobulin
  Arms: BUCY2

SUMMARY:
According to the 2022 ELN guidelines patients with high-risk acute myeloid leukemia were randomly divided into MA-BUCY2 conditioning group and BuCy2 conditioning group，to evaluate the efficacy and safety of two conditioning regimens in haploidentical hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
High risk acute myeloid leukemia patients were randomly divided into two groups before conditioning of haploidentical hematopoietic stem cell transplantation.The control group will use the BUCY2 conditioning，and the experimental group will use mitoxantrone liposome combined with BUCY2 for conditioning. After transplantation，we will observe the difference of one year relapse rates between two goups，also the adverse reactions of conditioning，GVHD，OS and PFS of the patients in two groups also been observed.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria of 2022 ELN guidelines for high-risk acute myeloid leukemia;
* Patients with allogeneic stem cell transplantation indications;
* Age 18-60 (including upper and lower limits) ;
* No gender limit;
* ECOG score 0~2 points;
* Flow MRD was negative before transplantation;
* The organ function level must meet the following requirements: a) Liver: aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 3 times the upper limit of normal value (ULN), Total bilirubin (TBIL) ≤ 1.5 × ULN； b) Kidney: blood creatinine ≤ 1.5 × ULN； c) Coagulation function: international normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN； d) Normal cardiac function: that is, the ECG is normal or abnormal without clinical significance, and the left ventricular ejection fraction (LVEF) is greater than 60 or myocardial zymogram CK-MB is normal, pro-BNP is less than 900 pg/ml;
* The results of serum pregnancy test of female subjects with reproductive ability must be negative before the first use of the test drug;

Exclusion Criteria:

* Previously received doxorubicin or other anthracycline drugs, and the total cumulative dose of doxorubicin was more than 360 mg/m2;
* Hypersensitivity to any study drug or its components;
* Cardiac function and disease meet one of the following conditions:

  1. Long QTc syndrome or QTc interval>480 ms;
  2. Complete left bundle branch block, II or III degree atrioventricular block;
  3. Serious and uncontrolled arrhythmia requiring drug treatment;
  4. American New York Heart Association rating ≥ III;
  5. Cardiac ejection fraction (LVEF) is less than 60%;
  6. History of myocardial infarction, unstable angina pectoris, severe unstable ventricular arrhythmia or He has any arrhythmia requiring treatment, clinical history of serious pericardial disease, or acute ischemia or activity ECG evidence of abnormal conduction system.;\
* Active infection of hepatitis B and hepatitis C;
* Human immunodeficiency virus (HIV) infection;
* Patients with other malignant tumors;
* Pregnant and lactating women and patients of childbearing age who are unwilling to take contraceptive measures;
* Have a history of abuse of drugs;
* History of mental illness or cognitive impairment; .Other researchers judged that it was not suitable for this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 264 (Estimated)
Dates: Start 2023-04-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
relapse rates | one year after transplantation
  blast cells in bone marrow are greater than or equal to 5%. Blast cells can be seen in peripheral blood or extramedullary relapse occurred.

SECONDARY OUTCOMES:
AEs | from beginning of the conditioning to one month after conditioning
  adverse reactions of conditioning regimen include nausea, vomiting, abdominal pain, diarrhea, heart, liver and kidney toxicity
aGVHD | At day 100 post-transplantation
  the incidence of acute graft versus host disease
OS | From date of diagnosis until the end of follow-up or the date of death from any cause, whichever came first，assessed up to 36 months.
  overall survival
PFS | From date of HSCT until the end of follow-up or the date of disease relapse from any cause, whichever came first，assessed up to 36 months.
  progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoning Wang, M.D., Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China